CLINICAL TRIAL: NCT01175928
Title: Phase 2 Study of the NormaTec PCD in the Treatment of Diabetic Peripheral Neuropathy
Brief Title: Pneumatic Medicine: A Transformative Treatment for Diabetic Peripheral Neuropathy
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: NormaTec Industries LP (Industry)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NormaTec_90513134-01; 1R43DK088634-01 (NIH)
Record Dates: First submitted 2010-08-03; First posted 2010-08-05 (Estimated); Last update posted 2012-04-20 (Estimated); Status verified 2012-04

CONDITIONS: Diabetic Polyneuropathy
Keywords: Diabetic polyneuropathy; Pneumatic Compression Device
MeSH Terms: conditions — Diabetic Neuropathies

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Peristaltic Pulse PCD (Experimental): Peristaltic Pulse Pneumatic Compression Device (NormaTec PCD)
  Interventions: Device: NormaTec PCD (Peristaltic Pulse PCD)
- Sham Device (Sham Comparator): Sham Pneumatic Compression Device (looks and sounds like real device, but applies no compression)
  Interventions: Device: Sham device

INTERVENTIONS:
Device: Sham device — Home treatment with PCD to both legs: 2 sessions of 1 hour duration every day
  Other Names: NormaTec PCD (sham device)
  Arms: Sham Device
Device: NormaTec PCD (Peristaltic Pulse PCD) — Home treatment with PCD to both legs: 2 sessions of 1 hour duration every day
  Other Names: NormaTec PCD
  Arms: Peristaltic Pulse PCD

SUMMARY:
The purpose of this study is to evaluate the efficacy of the NormaTec PCD, a non-invasive pneumatic compression device with the patented peristaltic pulse pneumatic waveform, in the treatment of Diabetic Peripheral Neuropathy (DPN).

The study will compare treatment with a NormaTec PCD and a sham device to assess whether the NormaTec PCD improves the signs and symptoms of DPN.

DETAILED DESCRIPTION:
Diabetes frequently leads to decreased sensation in the legs caused by diabetic peripheral neuropathy (DPN). DPN is an important risk factor for the development of foot ulceration, one of the most common causes for hospital admissions and lower-limb amputations among diabetic patients. However, to date there are no medications currently approved by the Food and Drug Administration to treat DPN.

The goal of this research project is to assess the effectiveness of a non-invasive, patented peristaltic pulse pneumatic compression device (the NormaTec PCD) in a home treatment program to improve the symptoms of DPN (e.g. numbness, pain, and tingling in the legs) and the underlying functioning of the nerves in the legs (as determined by sensory perception assessments and Nerve Conduction Studies testing).

In this prospective, randomized, double-blind study, subjects will be randomly placed in one of two groups: a control group using a sham NormaTec PCD ("placebo"); and an experimental group using a NormaTec PCD.

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed with type 1 or type 2 diabetes
* Patient diagnosed with distal symmetric polyneuropathy (DPN) attributable to diabetes
* A1C ≤ 11%
* Abnormal peroneal motor nerve conduction study where CMAP amplitude is less than 4 mV bilaterally.

Exclusion Criteria:

* Refuses consent
* Unlikely to be compliant with the research protocol as judged by the clinical investigator
* Neuropathy documented to be caused by something other than diabetes
* Medication for neuropathic pain initiated within the previous 3 months (to avoid confounding the results of the study)
* Medication for glucose control changed within the previous 3 months (to avoid confounding the results of the study)
* Documented DVT within the previous 3 months (since an acute DVT is a contraindication for Pneumatic Medicine treatment)
* Significant hepatic disease as judged by the clinical investigator (that might cause neuropathy unrelated to diabetes)
* Documented cancer treatment within the past 5 years (that might cause neuropathy unrelated to diabetes)
* History of exposure to neurotoxins or heavy metals (that might cause neuropathy unrelated to diabetes)
* Documented alcohol or drug abuse (that might cause neuropathy unrelated to diabetes)
* Documented major psychiatric disorder (that could contribute to non-adherence to the protocol)
* Presence of a major lower extremity amputation (since unable to perform bilateral distal sensory perception testing of the feet and NCS on the peroneal motor nerve)
* Significant peripheral arterial disease defined as an ankle-brachial index ("ABI") < 0.6 (to avoid critical limb ischemia and thus the high likelihood of the patient requiring a major amputation in the near future with drop out from the study)
* Severe lower extremity edema as judged by the clinical investigator (in order to not confound the results)
* End stage DPN where the peroneal motor nerve conduction results of both legs show an Amplitude = 0 mV
* Currently participating in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-10; Primary Completion 2012-09 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
Nerve Conduction Studies | 3 months
  Nerve conduction studies of the peroneal motor nerve performed bilaterally (amplitude, velocity, distal latency).
Nerve Conduction Studies | 1 month
  Nerve conduction studies of the peroneal motor nerve performed bilaterally (amplitude, velocity, distal latency).
Nerve Conduction Studies | 2 months
  Nerve conduction studies of the peroneal motor nerve performed bilaterally (amplitude, velocity, distal latency).

SECONDARY OUTCOMES:
Sensory perception measurements | baseline; 1 month; 2 months; 3 months
  Non-invasive sensory perception will be assessed with a 10-g monofilament (pressure); a 128 Hz tuning fork and a Neurothesiometer (vibration); a toothpick (sharp sensation); a cotton ball (soft sensation); an iced tuning fork (cold sensation); and calculation of the Neuropathy Disability Score.
Quality of life questionnaires | baseline; 1 month; 2 months; 3 months
  The following questionnaires will be self-administered: Norfolk Quality-of-Life Questionnaire for Diabetic Neuropathy (QOL-DN); Neuropathy Total Symptom Score-6 (NTSS-6); Problem Areas in Diabetes (PAID)

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Spirito, MD, Principal Investigator — Saints Medical Center
Locations (1):
- NormaTec, Newton Center, Massachusetts, United States